CLINICAL TRIAL: NCT02156908
Title: D-serine and Cognitive Remediation in Schizophrenia: Open Label Pilot
Brief Title: D-serine and Cognitive Remediation in Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nathan Kline Institute for Psychiatric Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 601945
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Schizophrenia
Keywords: cognitive remediation
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- D-serine (Experimental): D-serine
  Interventions: Drug: D-serine

INTERVENTIONS:
Drug: D-serine — D-serine 60 mg/kg

SUMMARY:
The investigators will test the effects of 3 days of D-serine (DSR) on auditory plasticity in a sensory based remediation (SBR) paradigm

DETAILED DESCRIPTION:
We will enroll 8 subjects in an open label, three session pilot in patients will receive three sessions of tone matching SBR.

5 Subjects will receive D-serine (60mg/kg) taken 1x each week during the SBR sessions. Subjects will receive study drug 30 minutes prior to session.

3 subjects received no intervention

ELIGIBILITY:
Inclusion criteria:

* 18 to 64 years old,
* IQ≥85 and
* estimated Glomerular Filtration Rate (GFR) ≥60. All oral and depot antipsychotics (with the exception of clozapine) are allowable. Patients must be on their antipsychotic medication for 1 month and stable on dose of antipsychotic and adjunctive medications for 2 weeks prior to study entry.

Exclusion criteria:

* history of neurological visual or hearing impairment,
* active suicidal ideation on the Columbia Suicide Severity Rating Scale (C-SSRS),
* current alcohol or drug abuse (<1 month) or substance dependence (<4 months). All women of child-bearing potential must have a negative urine pregnancy test at the baseline visit. We require an IQ of ≥85 to ensure that subjects will have a capacity to learn. In our cross-sectional studies, we have observed an IQ≥85 in over 90% of candidates, suggesting that this is not an overly restrictive criterion.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua T Kantrowitz, MD, Principal Investigator — Nathan Kline Institute
Locations (1):
- Nathan Kline Institute, Orangeburg, New York, United States

REFERENCES:
- [Result] Kantrowitz JT, Epstein ML, Beggel O, Rohrig S, Lehrfeld JM, Revheim N, Lehrfeld NP, Reep J, Parker E, Silipo G, Ahissar M, Javitt DC. Neurophysiological mechanisms of cortical plasticity impairments in schizophrenia and modulation by the NMDA receptor agonist D-serine. Brain. 2016 Dec;139(Pt 12):3281-3295. doi: 10.1093/brain/aww262. PMID 27913408

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Please see NCT01474395 for a related parallel study involving 13 schizophrenia patients and 13 healthy controls. Participants in NCT01474395 were not enrolled in the current study, i.e., both studies included separate groups of participants
Groups:
- D-serine: D-serine
  D-serine: D-serine 60 mg/kg (3 sessions, open label)
- No Intervention: 3 sessions without D-serine
Period: Overall Study
Arm/Group | D-serine | No Intervention
Started | 5 | 3
Completed | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D-serine | No Intervention | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (9.4) | 45.4 (14.3) | 44.0 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Mismatch Negativity (MMN)
Description: An MMN event is evoked by a discernible change in the pitch of a repetitive auditory stimulation. The stronger the response to a difference (i.e., the more negative the amplitude of the MMN), the better the outcome.
  MMN was obtained to pitch deviant stimuli pre-post auditory plasticity training, utilizing deviants to the same base frequencies as the auditory plasticity sessions, (i.e. 500, 1000, and 2000 Hz), with ~10 minutes of each base frequency. MMN will be conducted at baseline and after the final session. Reported outcome is change in MMN between baseline and final within session.
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: micro volts
Arm/Group | D-serine | no Intervention
Number analyzed (Participants) | 5 | 3
micro volts | .086 (0.36) | 0.31 (.29)

2. Secondary Outcome: Tone Matching Threshold
Description: Change tone matching threshold (the percent difference in pitch of two consecutively played tones that can be distinguished), higher numbers represent better outcomes. D-serine outcomes are for 2 consecutive D-serine sessions
Time Frame: three weeks
Measure: Mean (Standard Deviation); unit: percentage of difference in pitch
Arm/Group | D-serine | No Intervention
Number analyzed (Participants) | 5 | 3
percentage of difference in pitch | 11 (3.6) | 2.3 (0.7)

ADVERSE EVENTS:
Time Frame: 3 weeks
Groups:
- no Intervention: no intervention
Arm/Group | D-serine | no Intervention
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 0/5 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes